CLINICAL TRIAL: NCT00730613
Title: Pilot Feasibility and Safety Study of Cellular Immunotherapy for Recurrent/Refractory Malignant Glioma Using Genetically-Modified Autologous CD8+ T Cell Clones
Brief Title: Cellular Adoptive Immunotherapy Using Genetically Modified T-Lymphocytes in Treating Patients With Recurrent or Refractory High-Grade Malignant Glioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01020; P30CA033572 (NIH); CHNMC-01020; CDR0000590506 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2008-08-07; First posted 2008-08-08 (Estimated); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult anaplastic astrocytoma; adult diffuse astrocytoma; adult pilocytic astrocytoma; adult subependymal giant cell astrocytoma; adult anaplastic ependymoma; adult ependymoma; adult myxopapillary ependymoma; adult subependymoma; adult anaplastic oligodendroglioma; adult oligodendroglioma; adult brain stem glioma; adult giant cell glioblastoma; adult glioblastoma; recurrent adult brain tumor; adult gliosarcoma; adult mixed glioma; adult pineal gland astrocytoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Astrocytoma; Ependymoma; Glioma, Subependymal; Oligodendroglioma; Glioblastoma; Brain Neoplasms; Gliosarcoma; Glioma | interventions — Gene Expression Profiling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (therapeutic autologous lymphocytes) (Experimental): Patients receive an infusion of autologous antigen-specific CD8+ cytotoxic T-lymphocyte clones over 5-10 minutes on days 1, 3, and 5 of weeks 1 and 2. Treatment repeats every 3 weeks for a total of 2 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: therapeutic autologous lymphocytes; Genetic: gene expression analysis; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: therapeutic autologous lymphocytes — Cycles of escalating cell dose infusions up to the target cell dose of 10(8)
Genetic: gene expression analysis — At the time of excess pathology samples documenting response/relapse
Other: laboratory biomarker analysis — CSF generated at the time of each T-cell dose

SUMMARY:
RATIONALE: Cellular adoptive immunotherapy may stimulate the immune system in different ways and stop cancer cells from growing.

PURPOSE: This clinical trial is studying the side effects of cellular adoptive immunotherapy using genetically modified T-lymphocytes and to see how well it works in treating patients with recurrent or refractory high-grade malignant glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the feasibility and safety of cellular immunotherapy utilizing ex vivo expanded autologous CD8-positive T-cell clones genetically modified to express the IL-13 zetakine chimeric immunoreceptor and the Hy/TK selection/suicide fusion protein in patients with recurrent or refractory, high-grade malignant glioma.

Secondary

* To evaluate the antitumor activity of adoptively transferred clones in these patients.
* To screen for the development of anti-IL13 zetakine and anti-HyTK immune responses in these patients.
* To evaluate the efficacy of ganciclovir administration for ablating transferred clones in vivo should toxicity be encountered.

OUTLINE:

* Leukapheresis and therapy preparation: Patients undergo leukapheresis to obtain peripheral blood mononuclear cells. T-cells isolated from the peripheral blood are then genetically modified, hygromycin-resistant cloned, expanded ex vivo, and cryopreserved until the first clinical or radiographic evidence of recurrence or progression. Patients with documented disease recurrence or progression undergo re-biopsy or re-resection of the tumor and placement of a reservoir-access device (Rickham shunt) into the tumor resection cavity prior to autologous T-cell clone infusion therapy.
* Autologous T-cell clone infusion: Patients receive an infusion of autologous antigen-specific CD8+ cytotoxic T-lymphocyte clones over 5-10 minutes on days 1, 3, and 5 of weeks 1 and 2. Treatment repeats every 3 weeks for a total of 2 courses in the absence of disease progression or unacceptable toxicity. Patients achieving tumor regression with residual disease by MRI after 4 courses of study therapy may receive up to 2 additional courses in the absence of disease progression, unacceptable toxicity, or a complete response.

Patients undergo blood, cerebrospinal fluid, and tissue sample collection periodically for correlative studies. Samples are assessed for IL13Rα2 expression levels, susceptibility to redirected T-cell effector mechanisms, and other tumor and T-cell activation markers.

After completion of study treatment, patients will be followed monthly for 3 months, then every 3 months for two years, and then annually for at least 15 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignant glioma at original diagnosis

  * Grade III or IV disease
  * Refractory or recurrent disease
  * Unifocal site of original disease in cerebral cortex
* No clinical evidence of progressive encephalopathy
* Has not undergone recent re-resection of recurrent or progressive disease
* No communication between the tumor resection cavity and the ventricles and deep cerebrospinal fluid pathways as documented by post-operative MRI scan

PATIENT CHARACTERISTICS:

* Karnofsky performance status 70-100%
* Life expectancy > 3 months
* WBC ≥ 2,000/dL
* ANC > 1,000/dL
* Platelet count ≥ 100,000/dL (unsupported by transfusion or growth factor)
* Creatinine < 1.6 mg/dL
* Bilirubin < 1.5
* SGOT and SGPT < 2 times upper limit of normal
* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception
* Able to understand protocol basic elements and/or risks/benefits of participating in this pilot study
* No requirement for supplemental oxygen to keep saturation > 95% that is not expected to resolve within 2 weeks
* No uncontrolled cardiac arrhythmia
* No hypotension requiring pressor support
* No renal dialysis dependency
* No refractory seizure disorder
* No concurrent non-malignant illness that is poorly controlled with treatment or is of such severity the investigators deem it unwise to enter the patient on protocol
* No severe infection for which patient is being treated
* No history of ganciclovir and/or Prohance contrast allergy or intolerance
* No HIV positivity within the past 3 months

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Must have recovered from major surgery
* At least 4 weeks since primary therapy and no steroid dependence
* At least 2 weeks since prior adjuvant cytotoxic chemotherapy and recovered
* No concurrent systemic corticosteroids, except for use in managing T-cell therapy toxicity
* No concurrent immunotherapy (i.e., interferons, vaccines, or other cellular products)
* No concurrent pentoxifylline
* No other concurrent investigative agents
* No concurrent ganciclovir or ganciclovir derivative
* No concurrent acyclovir for non-life threatening herpes virus infection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2002-02; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Feasibility | 1 year after the end of treatment on study
Safety | 1 year after the end of treatment on study

SECONDARY OUTCOMES:
Anti-tumor activity of adoptively transferred clones | 1 year after the end of treatment on study
Anti-IL 13 zetakine and anti-HyTK immune response in patients | 1 year after the end of treatment on study
Efficacy of ganciclovir for clone ablation (in the event of toxicity) | 1 year after the end of treatment on study

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Forman, MD, Principal Investigator — City of Hope Comprehensive Cancer Center